CLINICAL TRIAL: NCT06100653
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of BCG for Therapeutic Use in Preventing Postoperative Recurrence of Non-muscular Invasive Bladder Cancer in People Aged 18 and Over
Brief Title: BCG for Therapeutic Use Phase I Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LKM-2023-BCG01
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Non-muscular Invasive Bladder Cancer
Keywords: Safety and Tolerability
MeSH Terms: interventions — Therapeutic Uses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCG for therapeutic use clinical trial group (Experimental): Ten patients with non-muscular invasive bladder cancer ≥14 days after surgery were included.
  Interventions: Drug: BCG for therapeutic use

INTERVENTIONS:
Drug: BCG for therapeutic use — The 10 patients were infused with BCG 120mg dissolved in 40 ~ 50 mL normal saline once a week for 6 times, then once every 2 weeks for 3 times, and then once a month (30 days) for 10 times, with a total of 19 times.

SUMMARY:
This clinical study adopted a single-arm, open, single-centertrial design. The purpose of this study was to evaluate the safety and tolerability, PK characteristics, shedding and immune response characteristics of BCG for therapeutic use developed by Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. in patients aged 18 and over after transethral resection of non-muscular invasive bladder cancer.

DETAILED DESCRIPTION:
This clinical study adopted a single-arm, open, single-centertrial design. The purpose of this study was to evaluate the safety and tolerability, PK characteristics, shedding and immune response characteristics of BCG for therapeutic use developed by Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. in patients aged 18 and over after transethral resection of non-muscular invasive bladder cancer.

This study includes three stages: screening period, observation period of administration, and safety follow-up period.

Screening period:

within 28 days before the first administration, the subjects will be eligible for enrollment confirmation.

Observation period of administration:

10 patients with non-muscular invasive bladder cancer ≥ 14 days after operation were included.The 10 patients were infused with BCG 120mg once a week for 6 times, then once every 2 weeks for 3 times, and then once a month (30 days) for 10 times, with a total of 19 times.

The peripheral blood samples of the subjects were collected to evaluate the exposure and immune response characteristics of the drugs in the blood, and the urine samples were collected to examine the immune response characteristics and shedding of the drugs. The safety data of each subject were observed ,collected and recorded, including vital signs, laboratory examination, adverse event (AE) and serious adverse event (SAE) (within 7 days after the first 5 times of each infusion treatment, and within 14 days after the sixth infusion (before V8 visit)). After 14 days of follow-up after the sixth infusion of the last subject, the clinical trial Data and Safety Monitoring Board (DSMB) will conduct an interim analysis to evaluate the safety and tolerability based on the obtained data. For the AE that did not recover within 14 days after the sixth infusion, the investigators should followe up until the AE was remission, or returned to the baseline, or the subject's condition was stable, or the subject lost follow-up / death.

When the subjects continued 13 times in the later period of bladder instillation therapy; blood routine examination was performed before the 10th, 13th, 16th and 19th instillation, and blood biochemical examination was performed before the 13th and 19th instillation. Cystoscopy and urine cytology were performed at the 3rd, 6th, 9th and 12th months after the first infusion. The subjects then continued their follow-up visits..

Safety follow-up period:

Safety follow-up was performed for7 days after the last administration. For the AE that did not recover 7 days after the last administration, the investigators should follow up to AE remission, or return to the baseline, or the subject's condition was stable, or the subject lost follow-up / death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and over after transurethral resection of non-muscular invasive bladder cancer, both male and female.

2. Voluntarily participate in the trial, provide valid identification, fully informed and signed a written informed consent form.

3. Eastern Cooperative Oncology Group (ECOG) score: 0 ~ 2. 4. According to the Guidelines for the Diagnosis and Treatment of Bladder Cancer (2022 edition), patients with histologically confirmed non-muscular invasive bladder cancer (NMIBC) who are assessed to be medium or high risk and need BCG intravesical instillation therapy (Patients who need secondary electroresection can be included in the study after the second electroresection is completed and the pathological results are confirmed to be medium-or high-risk non-muscular invasive bladder cancer). Excluding carcinoma in situ.

5. Clinical laboratory tests meet the following characteristics:

1. Blood routine: no hematopoietic growth factor or transfusion support was used within 14 days before enrollment, including absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5×109/L; Platelet ≥100000/mm3 or 100×109/L; Hemoglobin ≥9 g/dL.
2. Liver function: total serum bilirubin ≤1.5× upper limit of normal (ULN), total serum bilirubin <3×ULN, aspartate and alanine aminotransferase (AST and ALT) ≤2.5×ULN in subjects with Gilbert syndrome.
3. Renal function: creatinine clearance ≥45 mL/min (estimated according to Cockcroft Gault formula) or serum creatinine ≤1.5×ULN.
4. Coagulation function: activated partial thromboplastin time (APTT) ≤1.5×ULN, International normalized ratio (INR) ≤1.5×ULN.

Exclusion Criteria:

1. Any of the following:

1. Those who have immunodeficiency or impairment (such as AIDS patients), who are using immunosuppressive drugs or radiotherapy that are likely to cause systemic BCG disease reaction.
2. Allergic to BCG vaccine and its excipients.
3. Patients with a history of severe adverse reactions to BCG vaccine such as BCG septicemia or systemic infection.
4. Patients with acute or chronic active hepatitis B [Hepatitis B Surface Antigen (HBsAg) positive and peripheral blood hepatitis B virus deoxyribonucleic acid (DNA) copy number ≥103/mL], hepatitis C virus (HCV) antibody positive (HCV copy number ≥103/mL), human immunodeficiency virus (HIV) antibody positive, syphilis specific antibody positive, C-TST test strongly positive, active tuberculosis, patients who are receiving anti-tuberculosis treatment, and other patients with fever or acute infectious diseases.
5. Patients with a history of serious diseases of cardiovascular, cerebrovascular, lung, liver, kidney and other important organs, or those with severe hypertension or diabetes that can not be controlled clinically judged by the investigators; Patients with symptomatic urinary tract infections.
6. New York Heart Association (NYHA) heart function grade ≥3. 2. Patients with tumors of other genitourinary system or other organs. 3. Patients with carcinoma in situ (Tis stage) or muscular invasive bladder urothelial carcinoma (T2 stage and above).

4. Received any BCG treatment for NMIBC within 2 years before enrollment. Or recurrence of NMIBC after BCG treatment at any time.

5. Patients who had received chemotherapy, radiotherapy or immunotherapy within 4 weeks before admission (except for immediate postoperative intravesical chemotherapy).

6. Pregnant or lactating women (currently breastfeeding or less than one year after delivery although there is no artificial breastfeeding), women of childbearing age who cannot guarantee effective contraception during the trial period, and plan to have a pregnancy plan within 6 months after the last dosing (Including the partner of the male subject).

7. It is known or suspected that bladder perforation or abnormal conditions such as prolonged operation time and massive bleeding occur during the operation.

8. The investigator judged that there was severe gross hematuria before enrollment, and suspected that the surgical wound had not healed or the urinary tract mucosa was damaged.

9. with cystitis or having received other intravesical drug therapy and severe bladder irritation,which was judged by the investigator to be expected to affect the evaluation of this study.

10. Complete bladder incontinence, defined as the use of more than 6 pads within 24 hours.

11. Participated in clinical trials of other drugs within 3 months before enrollment.

12. Regular drinkers within six months before enrollment, such as those who drink more than 14 units of alcohol per week (1 unit =360 mL beer with 5% alcohol, or 45 mL spirits with 40% alcohol, or 150 mL wine with 12% alcohol); Or have a history of drug abuse or drug use.

13. The investigator believes that there may be any conditions that increase the risk of the subjects or interfere with the execution of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BCG for therapeutic use by medical examination, laboratory examination and follow-up | About 18 months through study completion, including observation period of administration and safety follow-up period
  1. After each infusion of the first 6 times:
     * Body temperature,
       * Blood pressure,
         * Pulse；
  2. Blood routine within 12 hours after each infusion of the first 6 times;
  3. Urine routine before each infusion for the first 6 times;
  4. On the 14th day after the 6th infusion (before administration of V8 visit):
     * Physiacl examination,
       * Vital signs,
         * Laboratory examination,
           * 12-lead ECG examination,
             * Color ultrasound of urinary system,
               * Imaging results ,
  5. All AE and SAE during 0-7 days after each infusion of the first 5 times;
  6. All AE and SAE within 14 days after the end of the 6th infusion ;
  7. During the 7th to 19th infusion of the experimental drug:
     * AE,
       * SAE ,
         * Tumor recurrence ,
  8. Examination results of safety follow-up : including AE, SAE, physical examination, vital signs, clinical laboratory examination , 12-lead ECG examination, color ultrasound of urinary system, imaging examination and so on.

SECONDARY OUTCOMES:
PK characteristics of BCG for therapeutic use by the level of Mycobacterium tuberculosis in the blood sample | 1h before the 1st and 6th administration and 2 h±30 min、24 h±2 h after the 1st and 6th administration
  The peripheral blood of the subjects was collected within 1h before the 1st and 6th administration and 2 h±30 min、24 h±2 h after the 1st and 6th administration to evaluate the exposure of BCG for therapeutic use in the blood.
  The levels of Mycobacterium tuberculosis (nucleic acid positive/negative) in the blood sample after the 1st and 6th administration were detected.
Immune response characteristics of BCG for therapeutic use by the level of cytokines in the blood and urine sample | before the 1st and 6th administration， 2 h±30 min and 24 h±2 h after the 1st and 6th administration， 2 h±1 h, 4 h±1 h, 8 h±2 h, and 24 h±3 h after 1st and 6th BCG administration .
  Blood sample collection: Peripheral blood samples of subjects were collected within 1 h before the 1st and 6th administration, and 2 h±30 min and 24 h±2 h after the 1st and 6th administration.
  Urine sample collection: last excreted urine of subjects were collected before the 1st and 6th administration, and excreted urine of subjects were collected 2 h±1 h, 4 h±1 h, 8 h±2 h, and 24 h±3 h after 1st and 6th BCG administration .
  The levels of interleukin 2 (IL-2), interleukin 6 (IL-6), interleukin 8 (IL-8), interleukin 12 (IL-12), interferon gamma (IFN- γ) and tumor necrosis factor (TNF) in blood and urine sample were detected.
Shedding of BCG for therapeutic use by the level of Mycobacterium tuberculosis in the urine sample | 1st and 3rd day after the 1st and 6th administration
  The urine excreted from the subjects were collected on the 1st and 3rd day after the 1st and 6th administration , in which the urine on the first day included 2 h ±1 h, 4 h ±1 h, 8 h ±2 h and 24 h ±3 h after BCG administration, and only once on the 3rd day to investigate the drug shedding.
  The levels of Mycobacterium tuberculosis (nucleic acid positive/negative) in the urine sample after the 1st and 6th administration were detected.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Sh Suan, Doctor, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, China

IPD SHARING:
Plan to Share IPD: No